CLINICAL TRIAL: NCT04338516
Title: Histological Evaluation of Healing Following Ridge Preservation Using a Composite Bovine Derived Xenograft or a Hydroxyapatite-Collagen Matrix
Brief Title: Ridge Preservation Using a Ossix™ Bone vs Bio-Oss® Collagen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Datum Dental LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC20190455H
Record Dates: First submitted 2020-04-05; First posted 2020-04-08 (Actual); Results first posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-11

CONDITIONS: TEETH EXTRACTION

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Bio-Oss® Collagen, (Active Comparator): subjects treated with Bio-Oss® Collagen, (Geistlich, Inc.)
  Interventions: Device: Bio-Oss® Collagen
- Ossix™ Bone (Experimental): subjects treated with Ossix™ Bone (Datum Dental Ltd)
  Interventions: Device: Ossix™ Bone

INTERVENTIONS:
Device: Ossix™ Bone — a resorbable sponge-like matrix of 80% hydroxyapatite and 20% sugar cross-linked porcine collagen
  Arms: Ossix™ Bone
Device: Bio-Oss® Collagen — 90% bovine derived xenograft granules and 10% porcine collagen
  Arms: Bio-Oss® Collagen,

SUMMARY:
This randomized, parallel design, controlled study will assess the histologic healing of this Ossix™ Bone in humans and compare it to a Bio-Oss® Collagen that is well researched.

Subjects will be enrolled into 2 groups. Each subject will provide a single non-molar tooth site for study treatment. The tooth will be extracted, the extraction socket will be filled with one of the study bone grafts. No wound dressing or membrane will be used to cover the bone graft material as both materials can be used alone. An core biopsy will be collected after 16 weeks of healing during the implant placement.

The study will evaluate if there is a difference in histologic wound healing following tooth extraction and ridge preservation between groups treated with Bio-Oss® Collagen compared to Ossix™ Bone.

ELIGIBILITY:
Inclusion Criteria:

* One tooth, excluding molars, that has been identified by dental faculty as requiring a single tooth extraction

  * A dental implant is indicated and treatment planned to replace the missing tooth
  * Have adequate restorative space for a dental implant-retained restoration
  * Have at least 10mm of alveolar bone height, without impinging on the maxillary sinus or inferior alveolar canal.
  * Have a dehiscence of the buccal or lingual bony plate of the tooth socket extending no more than 50% of the total depth of the socket.
  * Female patients who have undergone a hysterectomy, tubal ligation, or menopause, and non-pregnant women of child-bearing potential.
  * Are nonsmokers or former smokers. Current smokers may be included if they smoke <10 cigarettes per day

Exclusion Criteria:

* Will not cooperate with the follow-up schedule. Patients will not be entered who are mentally incompetent, prisoners, or pregnant.

  * Pregnant women or women intending to become pregnant during the study period (as confirmed verbally; an over the counter pregnancy test will be provided if pregnancy status is unknown or suspected).
  * Patients who become pregnant during the study will be withdrawn and standard care will be delivered.
  * Smokers who smoke >10 cigarettes per day
  * Clinical and/or radiographic determinations which will preclude inclusion in this study are: Active infection other than periodontitis; Inadequate bone dimensions or restorative space for a dental implant; Presence of a disease entity, condition or therapeutic regimen which decreases probability of soft tissue and bony healing, e.g., poorly controlled diabetes, chemotherapeutic and immunosuppressive agents, autoimmune diseases, history of bisphosphonate use or long-term steroid therapy; Positive medical history of endocarditis following oral or dental surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-03-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UT Health San Antonio (UTHSA), San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Casarez-Quintana A, Mealey BL, Kotsakis G, Palaiologou A. Comparing the histological assessment following ridge preservation using a composite bovine-derived xenograft versus an alloplast hydroxyapatite-sugar cross-linked collagen matrix. J Periodontol. 2022 Nov;93(11):1691-1700. doi: 10.1002/JPER.22-0149. Epub 2022 Jul 1. PMID 35661358

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bio-Oss® Collagen, | Ossix™ Bone
Started | 27 | 27
Completed | 23 | 21
Not Completed | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- BioOss Collagen; Ossix™ Bone: no adverse events were observed
- Total: Total of all reporting groups
Arm/Group | BioOss Collagen | Ossix™ Bone | Total
Number analyzed (Participants) | 27 | 27 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 27 | 54
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: YEARS] | 55 [27 to 80] | 55 [27 to 80] | 55 [27 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 14 | 14 | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 27 | 27 | 54

OUTCOME MEASURES:

1. Primary Outcome: Percent Vital Bone Formation,
Description: shows the amount of new bone formed after the procedure
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: percentage of vital bone
Arm/Group | Bio-Oss® Collagen, | Ossix™ Bone
Number analyzed (Participants) | 23 | 21
percentage of vital bone | 26.8 (15.8) | 39.3 (17.8)

2. Primary Outcome: Percent Residual Graft Material
Description: shows how much of the graft material remained intact
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: percentage of residual graft
Arm/Group | Bio-Oss® Collagen, | Ossix™ Bone
Number analyzed (Participants) | 23 | 21
percentage of residual graft | 17.9 (13.6) | 0 (0)

3. Primary Outcome: Percent Fibrous Tissue and Marrow Space
Description: amount of tissue that is neither native bone or graft material
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: percentage of marrow
Arm/Group | Bio-Oss® Collagen, | Ossix™ Bone
Number analyzed (Participants) | 23 | 21
percentage of marrow | 55.2 (12.7) | 60.7 (17.8)

ADVERSE EVENTS:
Time Frame: 16 weeks
Groups:
- OSSIX™ Bone: no subject suffered any adverse event due to the materials tested
Arm/Group | BioOss Collagen | OSSIX™ Bone
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/21
Other Adverse Events (participants affected / at risk) | 0/23 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-24): https://cdn.clinicaltrials.gov/large-docs/16/NCT04338516/Prot_SAP_000.pdf